CLINICAL TRIAL: NCT03501667
Title: Boston Children's Hospital
Brief Title: Testing Pediatric Rheumatology Diagnostic Decision Support in Clinical Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Amir Kimia, MD, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IRB-P00027105
Record Dates: First submitted 2018-04-04; First posted 2018-04-18 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Pediatric Rheumatological Condition (i.e., Arthritis, SLE, Kawasaki's Disaese)
MeSH Terms: conditions — Arthritis; Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: Comparing use of deision support group (intervention group) to use of common literature (control group) among pediatric trainees treating patients with possible rheumatologic disorder
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data collected by an RA, PI and outcome assessment (I.e., data analyst) are blinded to which arm the participant was assigned to. Given use of software, the participant cannot be blinded to the arm he/she was assigned
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of decision support tool (Active Comparator): Trainee using decision support tool while assessing a clinical case. This intervention will affect the study participant fund of knowledge on the case.
  Interventions: Other: Use of decision support tool
- Use of UpToDate (Active Comparator): Control group, participants using current literature prior to assessing a clinical case. Allowing 10 minutes to read on a topic during clinical care is an active intervention in the study participant fund of knowledge.
  Interventions: Other: Use of UpToDate

INTERVENTIONS:
Other: Use of decision support tool — use of a decision support software during clinical assessment of a case
  Other Names: Use of SimulConsult
  Arms: Use of decision support tool
Other: Use of UpToDate — Control group, participants using current literature prior to assessing a clinical case. Allowing 10 minutes to read on a topic during clinical care is an active intervention in the study participant fund of knowledge.
  Other Names: Use of current literature
  Arms: Use of UpToDate

SUMMARY:
Boston Children's Hospital resources include SimulConsult which is a decision support tool available for use of BCH provider through the library portal. It is offered along other resources on that webpage (UpToDate, Micromedex, and VisualDx). See addendum 1.

Recently, a pediatric rheumatology arm was added to the expertise of SimulConsult, guided by our co-PI, Dr. Robert Sundel. As this tool is being offered and used, the investigators would like to assess metric of performance of this tool in enhancing participant trainees knowledge about the work up of patients with a potential rheumatologic disorder. See also www.ncbi.nlm.gov/pubmed/27964737 The investigators are conducting a clinical research to assess improvement in the clinical performance of study participants evaluating patients with a potential rheumatologic disorder. The intervention involved in using a computerized decision support tool already available in the Boston Children's Hospital domain. The outcome will be comparing this performance to that of an attending physician as the gold standard. We will assess the study participants performance across two locations: Emergency Department and Rheumatology clinic. Care to patients remains unchanged, as the workup plan and care is provided by an attending across both domains.

The investigators main hypothesis is that using a decision support tool will result in a higher agreement rate between study participants' differential diagnosis and work up plan compared with the gold standard (attending differential diagnosis and research plan).

DETAILED DESCRIPTION:
Boston Children's Hospital resources include SimulConsult which is a decision support tool available for use of BCH provider through the library portal. It is offered along other resources on that webpage (UpToDate, Micromedex, and VisualDx). See addendum 1.

Recently, a pediatric rheumatology arm was added to the expertise of SimulConsult, guided by our co-PI, Dr. Robert Sundel. As this tool is being offered and used, the investigators would like to assess metric of performance of this tool in enhancing study participants (trainees) knowledge about the work up of patients with a potential rheumatologic disorder. See also www.ncbi.nlm.gov/pubmed/27964737 The investigators are conducting a clinical research to assess improvement in the clinical performance of trainees evaluating patients with a potential rheumatologic disorder. The intervention involved in using a computerized decision support tool already available in the Boston Children's Hospital domain. The outcome will be comparing this performance to that of an attending physician as the gold standard. The investigators will assess the study participants performance across two locations: Emergency Department and Rheumatology clinic. Care to patients remains unchanged, as the workup plan and care is provided by an attending across both domains.

Our main hypothesis is that using a decision support tool will result in a higher agreement rate between study participants' differential diagnosis and work up plan compared with the gold standard (attending differential diagnosis and research plan).

ELIGIBILITY:
Inclusion Criteria:

A trainee at Boston Children's residency program (pediatrics, emergency medicine, pediatric emergency medicine, pediatric rheumatology)

Exclusion Criteria:

Opting out of the study (optional at any stage)

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparing DDx with that of the attending physician (gold standard) | through study completion, an average of 1 year
  Comparing DDx provided by the trainee with that of the attending physician (gold standard)
Comparing evaluation plan with that of the attending physician (gold standard) | through study completion, an average of 1 year
  Comparing evaluation plan laid out by the trainee with that of the attending physician (gold standard)

CONTACTS AND LOCATIONS:
Overall Officials: Amir A Kimia, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Segal MM, Athreya B, Son MB, Tirosh I, Hausmann JS, Ang EY, Zurakowski D, Feldman LK, Sundel RP. Evidence-based decision support for pediatric rheumatology reduces diagnostic errors. Pediatr Rheumatol Online J. 2016 Dec 13;14(1):67. doi: 10.1186/s12969-016-0127-z. PMID 27964737